CLINICAL TRIAL: NCT00554216
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Determine the Safety and Efficacy of VI-0521 in the Treatment of Obesity in an Adult Population With BMI ≥ 35
Brief Title: Study of VI-0521 Compared to Placebo in Treatment of Obesity in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OB-302
Record Dates: First submitted 2007-11-03; First posted 2007-11-06 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Obesity
Keywords: Obesity, morbid obesity
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VI-0521 Low (Experimental): VI-0521; low dose phentermine/topiramate (PHEN/TPM 3.75 mg/23 mg)
  Interventions: Drug: VI-0521
- VI-0521 Top (Experimental): Top Dose VI-0521 consisting of 15 mg of Phentermine and 92 mg of Topiramate.
  Interventions: Drug: VI-0521
- Placebo (Placebo Comparator): Placebo to match
  Interventions: Drug: Placebo matched phentermine/topiramate

INTERVENTIONS:
Drug: VI-0521 — 3.75 mg phentermine/23 mg topiramate
  Arms: VI-0521 Low
Drug: VI-0521 — 15 mg phentermine/92 mg topiramate
  Arms: VI-0521 Top
Drug: Placebo matched phentermine/topiramate — Placebo matched phentermine/topiramate
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two doses of VI-0521 compared to placebo in treatment of obesity in an adult population with BMI ≥ 35.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 35 kg/m2
* Informed consent
* 70 years of age or less
* Triglyceride level ≤ 200 mg/dL with treatment of 0 or 1 medications
* Blood pressure of ≤ 140/90 mmHg with treatment of 0-2 medications for hypertension
* Fasting blood glucose level of ≤ 110 mg/dL

Exclusion Criteria:

* Stroke/myocardial infarction (MI)/unstable cardiovascular disease within 6 months
* Clinically significant renal, hepatic or psychiatric disease
* Unstable thyroid disease or replacement therapy
* Nephrolithiasis
* Obesity of known genetic or endocrine origin
* Participation in a formal weight loss program or lifestyle intervention
* History of glaucoma or intraocular pressure
* Pregnancy or breastfeeding
* Alcohol abuse
* Smoking cessation within previous 3 months or plans to quit smoking during study
* Eating disorders
* Cholelithiasis within past 6 months
* Excluded medications
* Type 2 diabetes
* Previous bariatric surgery
* History of bipolar disorder or psychosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1267 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peterson, Study Director — VIVUS LLC; Kishore Gadde, MD, Study Chair — Duke University
Locations (5):
- United States (5):
  - Research Site, San Diego, California
  - Research, Ridgefield, Connecticut
  - Research Site, Durham, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Austin, Texas

REFERENCES:
- [Derived] Guo F, Garvey WT. Cardiometabolic Disease Staging Predicts Effectiveness of Weight-Loss Therapy to Prevent Type 2 Diabetes: Pooled Results From Phase III Clinical Trials Assessing Phentermine/Topiramate Extended Release. Diabetes Care. 2017 Jul;40(7):856-862. doi: 10.2337/dc17-0088. Epub 2017 Apr 28. PMID 28455281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative sites in the US between November 2007 through May 2008
Groups:
- VI-0521 Low: PHEN/TPM 3.75 mg/23 mg
- VI-0521 Top: PHEN/TPM 15 mg/92 mg
Period: Overall Study
Arm/Group | Placebo | VI-0521 Low | VI-0521 Top
Started | 514 | 241 | 512
Completed | 272 | 147 | 340
Not Completed | 242 | 94 | 172
Not completed — Lost to Follow-up | 92 | 31 | 63
Not completed — Adverse Event | 16 | 16 | 36
Not completed — Withdrawal by Subject | 92 | 31 | 43
Not completed — Non compliance | 10 | 4 | 5
Not completed — Pregnancy | 2 | 1 | 14
Not completed — Restricted med | 3 | 1 | 1
Not completed — Other | 12 | 7 | 10
Not completed — Lack of Efficacy | 15 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- VI-0521 Low: PHEN/TPM 3.75/23
- VI-0521 Top: PHEN/TPM 15/92
- Total: Total of all reporting groups
Arm/Group | Placebo | VI-0521 Low | VI-0521 Top | Total
Number analyzed (Participants) | 514 | 241 | 512 | 1267
Age Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.76) | 43.0 (10.96) | 42.0 (12.21) | 42.6 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 425 | 201 | 424 | 1050
  Male | 89 | 40 | 88 | 217
Region of Enrollment [Number; unit: participants]
  United States | 514 | 241 | 512 | 1267

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Loss From Baseline to Week 56
Time Frame: baseline to 56 weeks
Population: intent-to-treat last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent weight loss
Arm/Group | Placebo | VI-0521 Low | VI-0521 Top
Number analyzed (Participants) | 498 | 234 | 498
percent weight loss | 1.55 (0.395) | 5.10 (0.538) | 10.92 (0.392)
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Top; With at least 250 subjects in each of the 3 arms in this trial, the trial has more than 90% power to detect a difference of at least 3.1% between combination and placebo treatment assuming a standard deviation of 5.3% and a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 9.36, 95% CI 2-sided [8.43 to 10.30], Standard Error of Mean 0.476
Statistical Analysis 2: Comparison: Placebo vs VI-0521 Low; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 3.54, 95% CI 2-sided [2.38 to 4.71], Standard Error of Mean 0.596
Statistical Analysis 3: Comparison: VI-0521 Low vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 5.82, 95% CI 2-sided [4.65 to 6.99], Standard Error of Mean 0.596

2. Primary Outcome: Percentage of Subjects With at Least 5% Weight Loss at Week 56
Time Frame: baseline to 56 weeks
Population: intent-to-treat last-observation-carried-forward (ITT-LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VI-0521 Low | VI-0521 Top
Number analyzed (Participants) | 498 | 234 | 498
percentage of participants | 17.3 | 44.9 | 66.7
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 9.61, 95% CI 2-sided [7.13 to 12.95], Standard Error of Mean 1.463
Statistical Analysis 2: Comparison: Placebo vs VI-0521 Low; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 3.97, 95% CI 2-sided [2.80 to 5.63], Standard Error of Mean 0.706
Statistical Analysis 3: Comparison: VI-0521 Low vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.76 to 3.33], Standard Error of Mean 0.394

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Description: Only subjects who received at least one dose of study drug were included in the safety analysis.
Arm/Group | Placebo | VI-0521 Low | VI-0521 Top
Serious Adverse Events (participants affected / at risk) | 14/513 | 6/240 | 13/511
Other Adverse Events (participants affected / at risk) | 374/513 | 192/240 | 432/511
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=513) | VI-0521 Low (N=240) | VI-0521 Top (N=511)
Cholelithiasis (Hepatobiliary disorders) | 3 | 1 | 1
Uterine Proplapse (Reproductive system and breast disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0
pancreatitus (Gastrointestinal disorders) | 1 | 0 | 0
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
hematuria (Renal and urinary disorders) | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0
angina pectoris (Cardiac disorders) | 1 | 0 | 0
hypertension (Vascular disorders) | 1 | 0 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
myocardial infarction (Cardiac disorders) | 0 | 1 | 0
cellulitis (Infections and infestations) | 0 | 1 | 0
appendicitis (Infections and infestations) | 0 | 1 | 0
thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
hypersensitivity (Immune system disorders) | 0 | 0 | 1
atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
staphylococcal infection (Infections and infestations) | 0 | 0 | 1
suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=513) | VI-0521 Low (N=240) | VI-0521 Top (N=511)
upper respiratory tract infection (Infections and infestations) | 56 | 38 | 63
nasopharyngitis (Infections and infestations) | 37 | 30 | 46
sinusitis (Infections and infestations) | 28 | 18 | 37
influenza (Infections and infestations) | 24 | 18 | 26
bronchitis (Infections and infestations) | 22 | 16 | 28
constipation (Gastrointestinal disorders) | 35 | 19 | 72
dry mouth (Gastrointestinal disorders) | 19 | 16 | 87
nausea (Gastrointestinal disorders) | 24 | 14 | 37
diarrhea (Gastrointestinal disorders) | 23 | 12 | 24
headache (Nervous system disorders) | 52 | 25 | 61
paresthesia (Nervous system disorders) | 10 | 10 | 96
dizziness (Nervous system disorders) | 21 | 7 | 29
dysgeusia (Nervous system disorders) | 5 | 3 | 43
back pain (Musculoskeletal and connective tissue disorders) | 26 | 13 | 28
insomnia (Psychiatric disorders) | 25 | 12 | 40
fatigue (General disorders) | 17 | 12 | 23
cough (Respiratory, thoracic and mediastinal disorders) | 18 | 8 | 26
vision blurred (Eye disorders) | 16 | 15 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.